CLINICAL TRIAL: NCT03829410
Title: A Phase 1b/2 Study of Onvansertib (PCM-075) in Combination With FOLFIRI and Bevacizumab for Second Line Treatment of Metastatic Colorectal Cancer in Patients With a KRAS Mutation
Brief Title: Onvansertib in Combination With FOLFIRI and Bevacizumab for Second Line Treatment of Metastatic Colorectal Cancer Patients With a KRAS Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TROV-054
Expanded Access: NCT04446793 (No longer available)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Colorectal Cancer; KRAS Gene Mutation
Keywords: KRAS mutation; PCM-075; Onvansertib; FOLFIRI; Irinotecan; 5-Fluorouracil; Leucovorin; Avastin; Bevacizumab; PLK1; PLK Inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — onvansertib; Bevacizumab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Onvansertib + FOLFIRI + Bevacizumab (Experimental): Phase 1b: Onvansertib escalating starting dose of 12 mg/m^2 orally Day 1 through Day 5 and Day 15 through Day 19 of each 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab. This Phase 1b portion of the study has been completed.
  Phase 2: Onvansertib Recommended Phase 2 Dose (RP2D) of 15 mg/m^2 orally Day 1 through Day 5 and Day 15 through Day 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab, with treatment modifications or delays based on unresolved toxicity experienced during a previous cycle.
  Interventions: Drug: Onvansertib; Biological: Bevacizumab; Drug: FOLFIRI

INTERVENTIONS:
Drug: Onvansertib — Onvansertib orally.
  Other Names: PCM-075
Biological: Bevacizumab — Bevacizumab intravenously.
  Other Names: Avastin®
Drug: FOLFIRI — FOLFIRI intravenously.

SUMMARY:
The purpose of the Phase 1b/2 study is to determine the safety and efficacy of Onvansertib, administered orally, daily on Day 1-5 and Day 15-19 of each 28-day cycle, in combination with FOLFIRI + Bevacizumab, as second-line treatment in adult participants who have metastatic colorectal cancer with a KRAS mutation. Participants must have histologically confirmed metastatic and unresectable disease, and previously failed treatment or be intolerant to fluoropyrimidine and oxaliplatin with or without bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic and unresectable colorectal cancer (CRC).
* Documentation of a KRAS mutation in exon 2, 3 or 4 in primary tumor or metastasis, assessed by a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. Participants with concomitant KRAS and BRAF-V600 mutations are excluded from this study. Participants with Microsatellite Instability High/Deficient Mismatch Repair (MSI-H/ddMMR) are also ineligible for enrollment in this study.
* Formalin-fixed, paraffin-embedded (FFPE) tumor tissue must be available for submission to a central laboratory in order for a participant to be eligible. If no archival tissue biopsy is available the participant must have a biopsy obtained at screening.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Signed informed consent for participation in the study.
* Participant is not receiving any other standard-of-care or experimental cancer therapy. Participants participating in non-interventional surveys or observational studies are allowed.
* Has failed treatment or is intolerant of fluoropyrimidine and oxaliplatin with or without bevacizumab.

  1. Participants must have had systemic therapy within 180 days of the screening visit, but can have no anti-cancer therapy within 28 days of the planned first day of treatment on study.
  2. Participants must have received oxaliplatin based chemotherapy with or without bevacizumab (>6 weeks in duration). Participants who received maintenance therapy with fluoropyrimidines are eligible with or without re-challenge with oxaliplatin in combination with fluoropyrimidines.
  3. Participants who received oxaliplatin/fluoropyrimidine-based neoadjuvant or adjuvant therapy and have disease recurrence or progression > 6 months from their last dose of neoadjuvant or adjuvant treatment (or > 6 months from surgery if no adjuvant therapy was administered) will be required to have received fluoropyrimidine/oxaliplatin-based therapy with or without bevacizumab as first-line treatment for metastatic disease.
  4. Participants must not have received prior irinotecan.
  5. For participants with rectal cancer, sequential neoadjuvant and adjuvant therapy will count as a single systemic regimen for advanced disease.
  6. Participants who discontinued first-line therapy because of toxicity are eligible for as long as progression occurred < 6 months after the last dose of first-line therapy.
* Chemotherapy regimen of irinotecan, fluorouracil [5-FU], and leucovorin (FOLFIRI) therapy is appropriate for the participant as determined by the Investigator.
* For a woman of child-bearing potential (WOCBP) or a male with a female partner who is a WOCBP: must have a negative serum or urine pregnancy test within 5 days prior to enrollment. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea > 12 consecutive months); or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device (IUD) or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child-bearing potential.
* Imaging computed tomography (CT)/ magnetic resonance imaging (MRI) of chest/abdomen/pelvis or other scans as necessary to document all sites of disease performed within 21 days prior to enrollment. Only participant with measurable disease as defined per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) are eligible for enrollment. CT is the preferred imaging modality, but MRI is also accepted.
* Must have acceptable organ function.
* Participant must consent to provision of, and Investigator(s) must confirm access to and agree to submit a representative, formalin fixed, paraffin block of tumor tissue to be used for correlative marker assays. Submission of the tissue does not have to occur prior to enrollment.
* Signed informed consent to provide blood sample(s) for specific correlative assays.

Exclusion Criteria:

* Concomitant KRAS and BRAF-V600 mutations or MSI-H/dMMR
* Anti-cancer chemotherapy or biologic therapy administered within 28 days prior to the first dose of study drug. The exception is a single dose of radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before randomization.
* More than one prior chemotherapy regimen administered in the metastatic setting.
* Major surgery within 6 weeks prior to enrollment.
* Untreated or symptomatic brain metastasis.
* Women who are pregnant or breastfeeding.
* Gastrointestinal (GI) disorder(s) that, in the opinion of the Investigator, would significantly impede the absorption of an oral agent (e.g., intestinal occlusion, active Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection).
* Unable or unwilling to swallow study drug.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure (CHF) Class II or higher according to the New York Heart Association (NYHA) Functional Classification, unstable angina pectoris, clinically significant cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.

  1. Known active infection with Human Immunodeficiency Virus (HIV), with measurable viral titer, and/or active infection with hepatitis B or C (participants who have had a hepatitis B virus [HBV] immunization are eligible).
  2. Known active infection with SARS-CoV-2.
  3. Clinically significant ascites or pleural effusions.
* Known hypersensitivity to 5-FU/leucovorin.
* Known hypersensitivity to irinotecan.
* Abnormal glucuronidation of bilirubin: known Gilbert's syndrome.
* Participants with a history of other malignancies except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix or prostate, or other solid tumors curatively treated with no evidence of disease for > 2 years.
* Any active disease condition that would render the protocol treatment dangerous or impair the ability of the participant to receive study drug.
* Planned concomitant use of medications known to prolong the QT/QTc interval according to institutional guidelines.
* Presence of risk factors for torsade de pointes, including family history of Long QT Syndrome or uncorrected hypokalemia.
* The following are exclusion criteria for bevacizumab:

  1. History of cardiac disease: CHF Class II or higher according to the New York Heart Association (NYHA); active coronary artery disease, myocardial infarction within 6 months prior to study entry; unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest) or cardiac arrhythmias requiring anti arrhythmic therapy (beta blockers or digoxin are permitted).
  2. Current uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management) and prior history of hypertensive crisis or hypertensive encephalopathy.
  3. History of arterial thrombotic or embolic events (within 6 months prior to study entry).
  4. Significant vascular disease (e.g., aortic aneurysm, aortic dissection, symptomatic peripheral vascular disease).
  5. Evidence of bleeding diathesis or clinically significant coagulopathy.
  6. Major surgical procedure (including open biopsy, significant traumatic injury, etc.) within 28 days, or anticipation of the need for major surgical procedure during the study, and minor surgical procedure (excluding placement of a vascular access device) within 7 days prior to study enrollment.
  7. Proteinuria at Screening as demonstrated by urinalysis with proteinuria ≥ 2+ (participants discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
  8. Abdominal fistula, GI perforation, peptic ulcer, or intra-abdominal abscess within the past 6 months.
  9. Ongoing serious, non-healing wound, ulcer, or bone fracture.
  10. Known hypersensitivity to any component of bevacizumab.
  11. History of reversible posterior leukoencephalopathy syndrome (RPLS).
* Use of strong CYP3A4 or UGT1A1 inhibitors or strong CYP3A4 inducers. Participants currently receiving these agents who are able to switch to alternate therapy are not excluded. Inhibitors should be stopped at least 1 week prior to the first dose of protocol therapy and inducers should be stopped at least 2 weeks prior to initiation of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - CARTI Cancer Center, Little Rock, Arkansas
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahn DH, Barzi A, Ridinger M, Samuelsz E, Subramanian RA, Croucher PJP, Smeal T, Kabbinavar FF, Lenz HJ. Onvansertib in Combination with FOLFIRI and Bevacizumab in Second-Line Treatment of KRAS-Mutant Metastatic Colorectal Cancer: A Phase Ib Clinical Study. Clin Cancer Res. 2024 May 15;30(10):2039-2047. doi: 10.1158/1078-0432.CCR-23-3053. PMID 38231047
- [Result] Ahn DH, Ridinger M, Cannon TL, Mendelsohn L, Starr JS, Hubbard JM, Kasi A, Barzi A, Samuelsz E, Karki A, Subramanian RA, Yemane D, Kim R, Wu CC, Croucher PJP, Smeal T, Kabbinavar FF, Lenz HJ. Onvansertib in Combination With Chemotherapy and Bevacizumab in Second-Line Treatment of KRAS-Mutant Metastatic Colorectal Cancer: A Single-Arm, Phase II Trial. J Clin Oncol. 2025 Mar;43(7):840-851. doi: 10.1200/JCO-24-01266. Epub 2024 Oct 30. PMID 39475591
- [Derived] Hagege A, Ambrosetti D, Boyer J, Bozec A, Doyen J, Chamorey E, He X, Bourget I, Rousset J, Saada E, Rastoin O, Parola J, Luciano F, Cao Y, Pages G, Dufies M. The Polo-like kinase 1 inhibitor onvansertib represents a relevant treatment for head and neck squamous cell carcinoma resistant to cisplatin and radiotherapy. Theranostics. 2021 Sep 21;11(19):9571-9586. doi: 10.7150/thno.61711. eCollection 2021. PMID 34646387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 68 participants from 7 investigative sites in the United States between June 2019 and January 2024.
Groups:
- Phase 1b: Onvansertib 12 mg/m^2: Oral onvansertib 12 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of each 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
- Phase 1b: Onvansertib 15 mg/m^2: Oral onvansertib 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of each 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
- Phase 1b: Onvansertib 18 mg/m^2: Oral onvansertib 18 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of each 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
- Phase 2: Onvansertib 15 mg/m^2: Oral onvansertib recommended phase 2 dose (RP2D) of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab, with treatment modifications or delays based on unresolved toxicity experienced during a previous cycle.
Period: Overall Study
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 | Phase 1b: Onvansertib 15 mg/m^2 | Phase 1b: Onvansertib 18 mg/m^2 | Phase 2: Onvansertib 15 mg/m^2
Started | 6 (Three participants enrolled in 15 mg/m^2 (2 in Phase 2 and 1 in Phase 1b) were inadvertently dosed at 12 mg/m^2.) | 8 (Three participants enrolled in 15 mg/m^2 (2 in Phase 2 and 1 in Phase 1b) were inadvertently dosed at 12 mg/m^2.) | 6 | 48 (Three participants enrolled in 15 mg/m^2 (2 in Phase 2 and 1 in Phase 1b) were inadvertently dosed at 12 mg/m^2.)
Completed | 0 | 0 | 0 | 1
Not Completed | 6 | 8 | 6 | 47
Not completed — Adverse Event | 1 | 0 | 1 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Disease Progressing | 3 | 4 | 2 | 31
Not completed — Miscellaneous | 2 | 4 | 3 | 10

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: defined as participants who received at least one dose of onvansertib in any cycle. Three participants enrolled in 15 mg/m^2 (2 in Phase 2 and 1 in Phase 1b) were inadvertently dosed at 12 mg/m^2 and are represented under Phase 1b 12 mg/m^2, as pre-specified in statistical analysis plan (SAP) section 9.4.
Groups:
- Phase 2: Onvansertib 15 mg/m^2: Oral onvansertib RP2D of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab, with treatment modifications or delays based on unresolved toxicity experienced during a previous cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 | Phase 1b: Onvansertib 15 mg/m^2 | Phase 1b: Onvansertib 18 mg/m^2 | Phase 2: Onvansertib 15 mg/m^2 | Total
Number analyzed (Participants) | 9 | 7 | 6 | 46 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.75) | 59.0 (14.39) | 57.5 (16.93) | 55.0 (9.82) | 56.3 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 3 | 19 | 31
  Male | 7 | 0 | 3 | 27 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 6 | 7
  Not Hispanic or Latino | 8 | 7 | 5 | 39 | 59
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 6 | 4 | 38 | 54
  Black or African American | 0 | 0 | 0 | 3 | 3
  Asian | 2 | 0 | 2 | 3 | 7
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Other | 1 | 0 | 0 | 1 | 2
  Not Reported | 0 | 0 | 0 | 1 | 1
Body Surface Area [Mean (Standard Deviation); unit: m^2] — BSA was calculated based on baseline weight and baseline height using the following formula: BSA (m^2) = 0.007184 * weight^0.425 * height^0.725.
  m^2 | 1.99 (0.315) | 1.82 (0.293) | 2.02 (0.316) | 1.97 (0.264) | 1.96 (0.277)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as a Grade 4 hematologic adverse events (AEs), Grade ≥ 3 non-hematologic AEs that were considered related to the study drug and that did not resolve within 14 days following presentation with standard management and care, Grade ≥ 3 thrombocytopenia with bleeding, neutropenic fever, any death not clearly due to the underlying disease or extraneous causes, or any change in liver function that met Hy's Law criteria of a DLT.
Time Frame: Up to Day 28
Population: Safety Analysis Set: defined as participants who received at least one dose of onvansertib in any cycle. Three participants enrolled in 15 mg/m^2 (2 in Phase 2 and 1 in Phase 1b) were inadvertently dosed at 12 mg/m^2 and are represented under Phase 1b 12 mg/m^2, as pre-specified in SAP section 9.4.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Onvansertib 12 mg/m^2: Oral onvansertib 12 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of each 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 | Phase 1b: Onvansertib 15 mg/m^2 | Phase 1b: Onvansertib 18 mg/m^2
Number analyzed (Participants) | 9 | 7 | 6
Participants | 1 | 1 | 3

2. Primary Outcome: Phase 1b: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: AEs were defined as any untoward medical occurrence associated with the use of a drug in humans. TEAEs are defined as any AE that started on or after the first day of study treatment and within 30 days of the last administration of study treatment, or that worsened on or after the first day of study treatment. AE severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 on a scale from Grade 1 (mild) to Grade 5 (death). An AE was considered "serious" if it resulted in death, life-threatening AE, hospitalization or prolongation of hospitalization, persistent or significant incapacity, or congenital anomaly/birth defect. The Investigator determined relatedness to the use of onvansertib.
  Clinically significant changes in vital signs, laboratory parameters, electrocardiograms, physical examinations, weight, and Eastern Cooperative Oncology Group (ECOG) performance status were reported as AEs.
Time Frame: Up to a maximum of 81 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 | Phase 1b: Onvansertib 15 mg/m^2 | Phase 1b: Onvansertib 18 mg/m^2
Number analyzed (Participants) | 9 | 7 | 6
Participants
  Any TEAE | 9 | 7 | 6
  Any TEAE Related to Onvansertib | 8 | 7 | 4
  Any TEAE CTCAE Grade ≥3 | 7 | 6 | 4
  Any TEAE CTCAE Grade ≥3 Related to Onvansertib | 4 | 1 | 1
  Any Serious TEAE | 2 | 3 | 1
  Any Serious TEAE Related to Onvansertib | 0 | 0 | 0

3. Primary Outcome: All-Treated Analysis Set: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants documented to have a confirmed complete response (CR) or partial response (PR) using the Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1). Two-sided 95% confidence interval (CI) was calculated using the exact binomial Clopper-Pearson method.
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: Up to a maximum of 131 weeks
Population: All-Treated Analysis Set: defined as participants who received at least 1 dose of assigned onvansertib in Cycle 1. Inclusive of the group of participants who were enrolled at 15 mg/m^2 in Phase 1b and Phase 2 (Part 1 and Part 2) as pre-specified in SAP section 9.4.2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2 Part 1: Onvansertib 15 mg/m^2: Oral onvansertib RP2D of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab, with treatment modifications or delays based on unresolved toxicity experienced during a previous cycle.
  Participants enrolled in Phase 2 before protocol v2 were categorized under Part 1 due to change in the Inclusion/Exclusion criteria.
- Phase 2 Part 2: Onvansertib 15 mg/m^2: Oral onvansertib RP2D of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab, with treatment modifications or delays based on unresolved toxicity experienced during a previous cycle.
  Participants enrolled in Phase 2 after protocol v2 were categorized under Part 2 due to change in the Inclusion/Exclusion criteria.
- Phase 1b and 2 Total: Onvansertib 15 mg/m^2: Oral onvansertib of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
Arm/Group | Phase 1b: Onvansertib 15 mg/m^2 | Phase 2 Part 1: Onvansertib 15 mg/m^2 | Phase 2 Part 2: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 33 | 13 | 53
percentage of participants | 42.9 [9.9 to 81.6] | 27.3 [13.3 to 45.5] | 15.4 [1.9 to 45.4] | 26.4 [15.3 to 40.3]

4. Secondary Outcome: Phase 2: Number of Participants With TEAEs
Description: AEs were defined as any untoward medical occurrence associated with the use of a drug in humans. TEAEs are defined as any AE that started on or after the first day of study treatment and within 30 days of the last administration of study treatment, or that worsened on or after the first day of study treatment. AE severity was graded according to the CTCAE version 5.0 on a scale from Grade 1 (mild) to Grade 5 (death). An AE was considered "serious" if it resulted in death, life-threatening AE, hospitalization or prolongation of hospitalization, persistent or significant incapacity, or congenital anomaly/birth defect. The Investigator determined relatedness to the use of onvansertib.
  Clinically significant changes in vital signs, laboratory parameters, electrocardiograms, physical examinations, weight, and ECOG performance status were reported as AEs.
Time Frame: Up to a maximum of 131 weeks
Population: Safety Analysis Set: defined as participants who received at least one dose of onvansertib in any cycle. Two participants from Phase 2 15 mg/m^2 were inadvertently dosed at 12 mg/m^2 dose level, as pre-specified in SAP section 9.4.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 46
Participants
  Any TEAE | 46
  Any TEAE Related to Onvansertib | 26
  Any TEAE CTCAE Grade ≥3 | 32
  Any TEAE CTCAE Grade ≥3 Related to Onvansertib | 8
  Any Serious TEAE | 17
  Any Serious TEAE Related to Onvansertib | 1

5. Secondary Outcome: All-Treated Analysis Set: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants documented to have a confirmed CR, PR or stable disease (SD) using the RECIST v1.1. Two-sided 95% CI was calculated using the exact binomial Clopper-Pearson method.
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: Up to a maximum of 131 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Onvansertib 15 mg/m^2 | Phase 2 Part 1: Onvansertib 15 mg/m^2 | Phase 2 Part 2: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 33 | 13 | 53
percentage of participants | 100 [59.0 to 100.0] | 90.9 [75.7 to 98.1] | 92.3 [64.0 to 99.8] | 92.5 [81.8 to 97.9]

6. Secondary Outcome: All-Treated Analysis Set: Progression-free Survival (PFS)
Description: PFS was defined as the time in months from the date of first administration of study treatment until the first observation of PD or death due to any cause, whichever occurs first, i.e.: (date of first PD or death date of first administration of study treatment +1)/30.4375. Median and 95% CI were calculated using the Kaplan-Meier method. Participants who did not have an observed documented PD or death from any cause were censored at the latest tumor response assessment date.
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: Up to a maximum of 131 weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Onvansertib 15 mg/m^2 | Phase 2 Part 1: Onvansertib 15 mg/m^2 | Phase 2 Part 2: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 33 | 13 | 53
months | 18 [3.7 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 6 [5.6 to 11.1] | 8 [3.9 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 8 [5.8 to 13.5]

7. Secondary Outcome: All-Treated Analysis Set: Duration of Response (DoR)
Description: DoR was calculated as the (date of first documented tumor progression or death due to any cause minus date of first documentation of a subsequently confirmed objective response plus 1)/30.4375. Participants who did not have an observed documented PD or death from any cause were censored at the latest tumor response assessment date.
Time Frame: Up to a maximum of 131 weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 1b and 2 Total: Onvansertib 15 mg/m^2: Oral onvansertib 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of each 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
Arm/Group | Phase 1b: Onvansertib 15 mg/m^2 | Phase 2 Part 1: Onvansertib 15 mg/m^2 | Phase 2 Part 2: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 33 | 13 | 53
months | 12 [NA to NA] — CIs were not calculable due to censoring and insufficient event data occurring near the median. | 12 [3.8 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | NA [NA to NA] — Median and CIs were not calculable as all participants were censored. | 12 [7.5 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median.

8. Secondary Outcome: All-Treated Analysis Set: Overall Survival (OS)
Description: OS was defined as the time in months from the date of first administration of study treatment until death due to any cause, i.e.: (Date of death date of first administration of study treatment +1)/30.4375. Participants who did not have documented death from any cause were censored at the date they were last known to be alive. OS was added as an endpoint with Protocol Amendment #1, therefore, OS data was only collected from then onward.
Time Frame: Up to a maximum of 131 weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Onvansertib 15 mg/m^2 | Phase 2 Part 1: Onvansertib 15 mg/m^2 | Phase 2 Part 2: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 33 | 13 | 53
months | NA [NA to NA] — Median and CIs were not calculable as all participants were censored. | NA [19.7 to NA] — Median and upper CI were not calculable due to fewer than 50% events. | NA [14.4 to NA] — Median and upper CI were not calculable due to fewer than 50% events. | NA [19.7 to NA] — Median and upper CI were not calculable due to fewer than 50% events.

9. Secondary Outcome: All-Treated Analysis Set: Percentage Change in KRAS-mutant Allelic Fraction (MAF)
Description: Blood samples were analyzed for the presence of circulating tumor DNA (ctDNA [including KRAS mutations]). KRAS-mutant allelic burden was based on liquid biopsies.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 (28-day cycle length)
Population: All-Treated Analysis Set: defined as participants who received at least 1 dose of assigned onvansertib in Cycle 1. Inclusive of the group of participants who were enrolled at 15 mg/m^2 in Phase 1b and Phase 2 (Part 1 and Part 2) as pre-specified in SAP section 9.4.2. Only participants with available data at Cycle 1 Day 1 and Cycle 2 Day 1 are represented.
Measure: Mean (Standard Deviation); unit: percentage change in MAF
Groups:
- Phase 1b: Onvansertib 15 mg/m^2; Phase 1b and 2 Total: Onvansertib 15 mg/m^2: Oral onvansertib of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
Arm/Group | Phase 1b: Onvansertib 15 mg/m^2 | Phase 2 Part 1: Onvansertib 15 mg/m^2 | Phase 2 Part 2: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 31 | 9 | 47
percentage change in MAF | -85.5857 (19.44200) | -76.2323 (26.43313) | -62.0000 (33.72414) | -74.9000 (27.45740)

10. Secondary Outcome: Phase 2: Observed Plasma Concentration at the End of Each Dosing Interval (Ctrough) of Onvansertib
Description: Plasma pharmacokinetic (PK) parameters for onvansertib were estimated using non-compartmental methods.
Time Frame: Pre-dose on Day 1 of Cycles 1 and 3 (28-day cycle length)
Population: PK Analysis Set: defined as all participants in the safety analysis set who had at least one evaluable plasma concentration of onvansertib.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 10
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6
  Cycle 1 Day 1 | 0.0000 (0.0000)
  Cycle 3 Day 1 | 0.3406 (0.34496)

11. Post Hoc Outcome: All-Treated Analysis Set: ORR by Bevacizumab Used in First-line Treatment
Description: ORR was defined as the percentage of participants documented to have a confirmed CR or PR using the RECIST v1.1. Two-sided 95% CI was calculated using the exact binomial Clopper-Pearson method. Data are presented by bevacizumab used in first-line treatment yes versus no.
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: Up to a maximum of 131 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1b; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2; Phase 1b; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2; Phase 1b and 2 Total; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2: Oral onvansertib 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of each 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
- Phase 2 Part 1; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2; Phase 2 Part 1; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2: Oral onvansertib RP2D of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab, with treatment modifications or delays based on unresolved toxicity experienced during a previous cycle.
  Participants enrolled in Phase 2 before protocol v2 were categorized under Part 1 due to change in the Inclusion/Exclusion criteria.
- Phase 2 Part 2; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2; Phase 2 Part 2; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2: Oral onvansertib RP2D of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab, with treatment modifications or delays based on unresolved toxicity experienced during a previous cycle.
  Participants enrolled in Phase 2 after protocol v2 were categorized under Part 2 due to change in the Inclusion/Exclusion criteria.
- Phase 1b and 2 Total; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2: Oral onvansertib of 15 mg/m^2 received on Days 1 through 5 and Days 15 through 19 of every 28-day cycle in combination with FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-FU, and 2400 mg/m^2 continuous intravenous infusion 5-FU + 5 mg/kg bevacizumab.
Arm/Group | Phase 1b; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 1b; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 1; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 1; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 2; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 2; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 0 | 22 | 11 | 11 | 2 | 40 | 13
percentage of participants | 42.9 [9.9 to 81.6] |  | 4.5 [0.1 to 22.8] | 72.7 [39.0 to 94.0] | 0 [0.0 to 28.5] | 100 [15.8 to 100.0] | 10.0 [2.8 to 23.7] | 76.9 [46.2 to 95.0]

12. Post Hoc Outcome: All-Treated Analysis Set: PFS by Bevacizumab Used in First-line Treatment
Description: PFS was defined as the time in months from the date of first administration of study treatment until the first observation of PD or death due to any cause, whichever occurs first, i.e.: (date of first PD or death date of first administration of study treatment +1)/30.4375. Median and 95% CI were calculated using the Kaplan-Meier method. Participants who did not have an observed documented PD or death from any cause were censored at the latest tumor response assessment date. Data are presented by bevacizumab used in first-line treatment yes versus no.
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: Up to a maximum of 131 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 1b; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 1; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 1; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 2; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 2 Part 2; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total; Bevacizumab Used in First-line Treatment: Onvansertib 15 mg/m^2 | Phase 1b and 2 Total; Bevacizumab Not Used in First-line Treatment: Onvansertib 15 mg/m^2
Number analyzed (Participants) | 7 | 0 | 22 | 11 | 11 | 2 | 40 | 13
percentage of participants | 18 [3.7 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. |  | 6 [3.6 to 6.1] | 15 [9.5 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 8 [3.7 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | NA [NA to NA] — Median and CIs were not calculable as all participants were censored. | 6 [5.3 to 8.4] | 15 [9.5 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median.

ADVERSE EVENTS:
Time Frame: Up to a maximum of 131 weeks
Description: Safety Analysis Set: defined as participants who received at least one dose of onvansertib in any cycle. Three participants enrolled in 15 mg/m^2 (2 in Phase 2 and 1 in Phase 1b) were inadvertently dosed at 12 mg/m^2 and are represented under Phase 1b 12 mg/m^2, as pre-specified in SAP section 9.4.
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 | Phase 1b: Onvansertib 15 mg/m^2 | Phase 1b: Onvansertib 18 mg/m^2 | Phase 2: Onvansertib 15 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7 | 0/6 | 1/46
Serious Adverse Events (participants affected / at risk) | 2/9 | 3/7 | 1/6 | 17/46
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7 | 6/6 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Onvansertib 12 mg/m^2 (N=9) | Phase 1b: Onvansertib 15 mg/m^2 (N=7) | Phase 1b: Onvansertib 18 mg/m^2 (N=6) | Phase 2: Onvansertib 15 mg/m^2 (N=46)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hepatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sigmoidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prolactin-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1b: Onvansertib 12 mg/m^2 (N=9) | Phase 1b: Onvansertib 15 mg/m^2 (N=7) | Phase 1b: Onvansertib 18 mg/m^2 (N=6) | Phase 2: Onvansertib 15 mg/m^2 (N=46)
Nausea (Gastrointestinal disorders) | 6 (9) | 6 (14) | 5 (9) | 29 (53)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 6 (13) | 3 (5) | 23 (61)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 6 (8) | 1 (1) | 18 (53)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 4 (11) | 3 (5) | 16 (20)
Vomiting (Gastrointestinal disorders) | 3 (11) | 4 (7) | 2 (2) | 11 (20)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (1) | 16 (21)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (6)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (6) | 0 (0) | 1 (3) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Gingival recession (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (22) | 7 (9) | 4 (8) | 36 (70)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (9)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 4 (7) | 3 (4) | 5 (12) | 18 (34)
White blood cell count decreased (Investigations) | 5 (10) | 2 (4) | 5 (9) | 13 (22)
Platelet count decreased (Investigations) | 4 (5) | 1 (1) | 3 (3) | 12 (22)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 1 (3) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 7 (11)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 6 (8)
Lymphocyte count decreased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 6 (18)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (11)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood chloride increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram ST-T segment abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wall motion score index abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 2 (2) | 4 (6) | 18 (29)
Neutropenia (Blood and lymphatic system disorders) | 2 (7) | 3 (5) | 2 (2) | 18 (38)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 4 (8)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 1 (1) | 10 (20)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 10 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (9)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 8 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 3 (3) | 14 (18)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (7) | 3 (3) | 2 (3) | 15 (42)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (5)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Lacrimation increased (Eye disorders) | 0/0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0/0 (0) | 0 (0) | 0 (0) | 1 (2)
Eye irritation (Eye disorders) | 0/0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental restoration failure (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Reaction to previous exposure to any vaccine (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (4)
Skin laceration (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site inflammation (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT03829410/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT03829410/SAP_001.pdf